CLINICAL TRIAL: NCT06599021
Title: Swallowing Difficulties in People Over 60 Years: Prevalence, Degree of Difficulty and Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Tuomi (Other)
Responsible Party: Sponsor-Investigator, Lisa Tuomi, Speech-language pathologist, associate professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00262-01
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Dysphagia; Intervention; Ageing
Keywords: Dysphagia; Age-related dysphagia; Health-related quality of life; Dysphagia intervention; Dysphagia characteristics
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscular strengthening training (Experimental): The muscular strengthening training is permformed 3 times daily as "head-ups" where the participant lies down and lifts their head anf then holds it upright during 60 seconds. This is repeated x 3 followed by 30 head-lifts. The duration of the training programme is 6 weeks.
  Interventions: Behavioral: Muscular strengthening training
- Skill-based training (Experimental): During the skill-based training programme, food and beverages are used as swallowing training material based on a pre-determined food-hierarchy. The training starts at the highest level that the participant can safely swallow and then progresses as strength and coordination of swallowing improves. This training is comprised of 15 speech- and language pathologist lead training sessions during 3 weeks.
  Interventions: Behavioral: Skill-based training
- Compensatory treatment (No Intervention): The control group will receive information about dysphagia and advise on compensatory strategies.

INTERVENTIONS:
Behavioral: Muscular strengthening training — 6 weeks daily muscular strengthening training.
  Arms: Muscular strengthening training
Behavioral: Skill-based training — 15 sessions skill based swallowing training lead by a speech and language pathologist during 3 weeks.
  Arms: Skill-based training

SUMMARY:
Participants included in SCAPIS2 (Swedish Cardio Pulmonary bioimage study) are screened regarding swallowing difficulty using a timed water swallow test. Participants who show signs of swallowing difficulty (dysphagia) are included in the present study, which encompasses s flexible endoscopic evaluation of swallowing function (FEES). Participants showing a moderate-severe dysphagia are randomized into one of three intervention groups: muscle strengthening training, skill-based swallowing training and a control group who will receive compensatory treatment. The study is expected to improve diagnostics and treatment of swallowing difficulties in an ageing population.

ELIGIBILITY:
Inclusion Criteria:

* Participation in SCAPIS2
* Swallowing dysfunction according to timed water swallow test or
* Swallowing dysfunction according to self-report

Exclusion Criteria:

* Severely impaired intellectual abilities.
* Inability to consent to inclusion in the study.
* Inability to answer written questionnaires in Swedish

Inclusion of non-dysphagia control cohort: No signs of aspiration, slow swallowing (<10 ml/sec) or self-rated difficulties with eating and swallowing in sub-study SCAPIS2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Penetration-aspiration score (PAS) | Baseline to post-intervention (6 weeks)
  Ranges from 1-8 where 8 indicates worst possible aspiration score. Swallowing safety measured from Flexible Endoscopic Examination of Swallowing (FEES).

SECONDARY OUTCOMES:
Dysphagia related symtoms | Up to 12 months post-intervention
  Patient reported outcome measurement (PROM) with Swallowing quality of life (Swal-QOL). Measures QOL depending of swallowing difficulty. Consists of 44 items divided into 10 domains and a symtom frequency scale. Scores on each domain is transformed into scores ranging from 0-100, where 100 indicates best possible swallowing QOL. The Swedish version has been fond valid and reliable.
Tongue strength | Up to 12 months post-intervention
  Anterior and posterior tongue strength during swallowing and maximal effort is measured with the Iowa Oral Performance Instrument (IOPI)
Body composition | Up to 12 months post-intervention
  Body composition will be measured using Bioelectric impedance analysis (BIA). Provides measures of fat-free mass and fat.
Cost of intervention | Up to 12 months post-intervention
  Will be provided through hospital records regarding number of hospital visits and in-hospital treatment during 1 year from start of intervention.
Self-perceived swallowing function | Up to 12 months post-intervention
  Measured with the Swedish Eating assessment tool (ÄT-10). 10 items with scores ranging from 0 to 40, higher scores indicates worse function. Scores above 3 points are considered to identify the prevalence of a swallowing dysfunction.
Quality of Life | Up to 12 months post-intervention
  Measured with the EuroQOL 5 domains (EQ5D). Each domain is rated on a scale from 1-3 where a higher number indicates lower QOL.
Quality of Life | Up to 12 months post-intervention
  Measured with the RAND-36. Scores range between 0-100, where 100 indicates best possible outcome.
Assessment of swallowing efficiency | Up to 12 months post-intervention
  Measurement of swallowing efficiency will be performed with the validated scale such as Yale oropharyngeal residue scale where scores range between 1-5 (none-severe)
Assessment of secretion | Up to 12 months post-intervention
  Measurement of swallowing function will be performed with assessment of secretion using a validated eight-point scale assesses secretion severity under the subcategories of location, amount, and response. Assessment is performed in a blinded manner.
Assessment of swallowing initiation | Up to 12 months post-intervention
  Initiation of swallowing will be assessed in a blinded manner, where initiation will be categorized referring to where te bolus reaches befor swallowing is initiated.
Assessment of overall swallowing function from the FEES | Up to 12 months post-intervention
  Measurement of swallowing function will be performed with the Swedish tool DIGEST-FEES (Dynamic Imaging Grade of Swallowing Toxicity; FEES = flexible endoscopic evaluation of swallowing). This be utilized to describe the severity of safety, efficiency, and pharyngeal stage overall swallowing impairment on FEES. The tool will be validated for the participant group through comparisons with the other measures of swallowing function. The scale ranges from 0 (normal) to 4=life threatening

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided